CLINICAL TRIAL: NCT00928889
Title: A Multi-center, Open-label, Randomized, Active-control, Parallel-group Designed Study to Compare Effects of Nateglinide and Acarbose on Postprandial Status in Chinese Drug-naive Type 2 Diabetes Mellitus Patients
Brief Title: Effects of Nateglinide vs Acarbose on Postprandial Glucose Fluctuation, Dyslipidemia, and Inflammatory Factors
Acronym: ENERGY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDJN608ACN06
Record Dates: First submitted 2009-06-25; First posted 2009-06-26 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes mellitus, type 2; nateglinide; acarbose; hyperglycemia; dyslipidemias; C-reactive protein
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Dyslipidemias | interventions — Nateglinide; Acarbose

ARMS (2):
- Nateglinide 120 mg (Experimental): Nateglinide was taken orally 3 times daily, 10 minutes before meals for 4 weeks.
  Interventions: Drug: Nateglinide 120 mg
- Acarbose 50 mg (Active Comparator): Acarbose 50 mg was taken orally 3 times daily, with the first bite of food at meals for 4 weeks.
  Interventions: Drug: Acarbose 50 mg

INTERVENTIONS:
Drug: Nateglinide 120 mg — Nateglinide 120 mg was supplied as tablets.
  Other Names: Starlix
  Arms: Nateglinide 120 mg
Drug: Acarbose 50 mg — Acarbose 50 mg was supplied as tablets.
  Other Names: Glucobay
  Arms: Acarbose 50 mg

SUMMARY:
This study was conducted to demonstrate superiority of nateglinide in postprandial glucose fluctuation, dyslipidemia, and inflammatory status improvement.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 2 diabetes mellitus patients
* HbA1c > 6.5 and < 9.0%
* Fasting fingertip capillary blood glucose (FCBG) < 9 mmol/L after 2 weeks diet control

Exclusion Criteria:

* History of acute metabolic complications in the past 3 months or of severe diabetic complications or severe infections or active substance abuse
* Liver disease
* Patients under oral hypoglycemic drugs and/or insulin treatment, or corticosteroid treatment within past 4 weeks

Other protocol-defined inclusion/exclusion criteria applied to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- China (6):
  - People's Liberation Army. The Military General Hospital of BeiJing, Beijing
  - Peiking University First Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - The First Affiliated Hospital, Zhongshan (Sun Yat-sen) University, Guangzhou
  - The Second Affiliated Hospital, Zhongshan (Sun Yat-sen) University, Guangzhou
  - Nanfang Hospital, the Affiliated South Hospital of the Southern Medical University, Guangzhou

REFERENCES:
- [Background] Gao HW, Xie C, Wang HN, Lin YJ, Hong TP. Beneficial metabolic effects of nateglinide versus acarbose in patients with newly-diagnosed type 2 diabetes. Acta Pharmacol Sin. 2007 Apr;28(4):534-9. doi: 10.1111/j.1745-7254.2007.00534.x. PMID 17376293

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Started | 80 | 80
Completed | 75 | 78
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg | Total
Number analyzed (Participants) | 80 | 80 | 160
Age Continuous [Mean (Standard Deviation); unit: years] | 53.1 (10.95) | 51.9 (10.82) | 52.5 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 33 | 73
  Male | 40 | 47 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Postprandial Glucose Excursion (PPGE) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of plasma glucose at 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. PPGE was defined as the mean difference between the preprandial glucose value and the postprandial glucose value measured at 2 hours in a standardized meal test. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM.
Time Frame: Baseline to the end of the study (Week 4)
Population: Intent-to treat population (ITT): All randomized participants who received at least 1 dose of study drug, had valid baseline data, and at least 1 post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L | -1.775 (1.3618) | -2.434 (1.4418)

2. Secondary Outcome: Change From Baseline in Peak Postprandial Glucose at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of plasma glucose at 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. The peak postprandial glucose values were used in the calculation of change from Baseline at Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L | -2.350 (1.8480) | -3.129 (1.8151)

3. Secondary Outcome: Change From Baseline in Postprandial Glucose Area Under the Curve at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of plasma glucose at 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. The postprandial glucose area under the curve was calculated using values from the 4 time points. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol*min/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol*min/L | -217.628 (179.8929) | -278.447 (171.2480)

4. Secondary Outcome: Change From Baseline in Total Cholesterol at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of total cholesterol prior to (fasting) and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. Total cholesterol was assessed at each study site using the same method and same reference value.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L
  Fasting, N=74, 77 | 0.015 (0.742) | -0.149 (1.050)
  120 minutes, N=74, 76 | 0.010 (0.700) | -0.059 (0.682)

5. Secondary Outcome: Change From Baseline in Triglycerides at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of triglycerides prior to (fasting) and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. Triglycerides were assessed at each study site using the same method and same reference value.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L
  Fasting, N=74, 77 | -0.010 (0.737) | -0.418 (1.047)
  120 minutes, N=74, 76 | 0.026 (0.676) | -0.396 (0.891)

6. Secondary Outcome: Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of LDL-C prior to (fasting) and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. LDL-C was assessed at each study site using the same method and same reference value.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L
  Fasting, N=74, 77 | 0.036 (0.634) | 0.036 (0.570)
  120 minutes, N=74, 76 | -0.000 (0.604) | 0.044 (0.589)

7. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of HDL-C prior to (fasting) and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. HDL-C was assessed at each study site using the same method and same reference value.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 74 | 77
mmol/L
  Fasting, N=74, 77 | 0.020 (0.150) | -0.039 (0.130)
  120 minutes, N=74, 76 | 0.023 (0.246) | 0.003 (0.276)

8. Secondary Outcome: Change From Baseline in Free Fatty Acids (FFA) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of FFA prior to (fasting) and 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. FFA was assayed at a central laboratory.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 73 | 75
mmol/L
  Fasting, N=73, 75 | -0.048 (0.251) | -0.040 (0.213)
  30 minutes, N=73, 75 | -0.112 (0.427) | -0.048 (0.363)
  60 minutes, N=72, 75 | -0.224 (0.482) | -0.048 (0.383)
  90 minutes, N=72, 75 | -0.109 (0.438) | -0.042 (0.419)
  120 minutes, N=73, 75 | -0.099 (0.605) | -0.034 (0.490)

9. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (hsCRP) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of hsCRP prior to (fasting) and 30, 60, 90, and 120 minutes following the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. hsCRP was assayed at a central laboratory.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 73 | 75
mg/dL
  Fasting, N=73, 75 | -0.229 (1.207) | 0.080 (0.404)
  30 minutes, N=73, 75 | -0.227 (1.232) | 0.024 (0.135)
  60 minutes, N=72, 75 | -0.219 (1.122) | 0.071 (0.398)
  90 minutes, N=72, 75 | -0.220 (1.231) | 0.077 (0.394)
  120 minutes, N=72, 74 | -0.218 (1.254) | 0.074 (0.375)

10. Secondary Outcome: Change From Baseline in Glycosylated Serum Albumin (GSA) at the End of the Study (Week 4)
Description: Blood samples were collected for measurement of GSA prior to (fasting) the start of a standardized meal test at Baseline and Week 4. Participants were fasting (no calorie intake for at least 8 hours prior to the meal test) and completed the standardized meal test between 7 and 10 AM. GSA was assayed at a central laboratory.
Time Frame: Baseline to the end of the study (Week 4)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Number analyzed (Participants) | 72 | 75
Percentage | -1.2 (1.57) | -1.2 (2.13)

ADVERSE EVENTS:
Time Frame: Baseline to the end of the study (Week 4)
Description: Safety Population.
Arm/Group | Nateglinide 120 mg | Acarbose 50 mg
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80
Other Adverse Events (participants affected / at risk) | 5/80 | 7/80
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nateglinide 120 mg (N=80) | Acarbose 50 mg (N=80)
Abdominal distension (Gastrointestinal disorders) | 1 | 4
Flatulence (Gastrointestinal disorders) | 1 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.